CLINICAL TRIAL: NCT03868878
Title: Twelve Weeks of Capoeira Training Decrease Plasma Triglycerides in Advanced-age Frail Adults of a Long-term Institution
Brief Title: Capoeira Training Decrease Plasma Triglycerides
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do vale do São Francisco (Other)
Collaborators: Regional Hospital of Juazeiro, BA, Brazil (Unknown); Fundação de Amparo à Ciência e Tecnologia de Pernambuco (Other)
Responsible Party: Principal Investigator, Sérgio Rodrigues Moreira, Professor (PhD), Universidade Federal do vale do São Francisco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3
Record Dates: First submitted 2019-03-05; First posted 2019-03-11 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Physical Conditioning, Human; Lipid Metabolism; Aged
Keywords: Capoeira Training (martial arts); Triglycerides; Aging
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Capoeira training group (Experimental): The experimental protocol for Capoeira program lasted 12 weeks and was performed twice a week with duration of 60 minutes each with warm-up, basic movements in the modality, and 20 minutes with theoretical instructions related to Capoeira and musicality.
  Interventions: Other: Capoeira training
- Control group (Sham Comparator): While the Capoeira group performed the entire class, the Control group performed only the final part (20 minutes) with musicality - singing and touch of typical instruments - and theoretical instructions related to Capoeira.
  Interventions: Other: Capoeira training

INTERVENTIONS:
Other: Capoeira training — The Capoeira training protocol, based in the modern styles was applied by an instructor with 16 years of experience. The protocol followed the directions of the ABADÁ Capoeira system, being adapted to the sample of older adults of the present study. The experimental protocol for Capoeira progressive training program lasted 12 weeks and was performed twice a week with duration of 60 minutes each. Each session was divided in three parts, being: 1) initial part: consisting of 10 minutes warm-up with recreational activities at low intensity; 2) main part: consisting of 30 minutes of basic movements in the modality and; 3) final part: consisting of 20 minutes with theoretical instructions related to Capoeira and musicality (singing and touch of typical instruments). In order to perform the Capoeira progressive training program, the technical improvement naturally occurred every week, resulting in a higher speed in movements execution and thus to a gradual increase in training intensity.
  Other Names: Physical training: attack / defense movements

SUMMARY:
Background: Among the risk factors associated with aging, a special highlight has been attributed to cardiovascular dysfunctions, insulin resistance, central obesity and dyslipidemia, which is marked by low levels of cholesterol (high density lipoprotein) and in particular by high levels of plasma triglycerides. Individuals with high levels of plasma triglycerides tend to have a prolonged postprandial hypertriglyceridemia after a fat-meal challenge, which would potentially further increase the risk associated with cardiovascular disease. Due to the impact of aging and its associated risk factors on the older adults health, several strategies have been proposed to avoid the progression of chronic diseases. These diseases are frequent in this population, especially the ones that resides in long-term institutions and they are mainly characterized by sedentary lifestyle and functional inability. Systematic reviews have shown that the implementation of physical activity programs associated with a favorable dietary pattern may benefit the lipid profile of the older adults. Moreover, it is suggested as a primary strategy, the realization of physical exercise as a therapy for this disease. In the physical exercise programs aspects, unconventional modalities such as Capoeira, which is practiced in more than 150 countries, it has aroused interest in the scientific research. Characterized by a system composed by attack and defense movements and from Afro-Brazilian origin, Capoeira combines sports elements of the fight, gymnastics, dance and musicality. However, there is no study investigating the effect of Capoeira training on the lipid profile of older adults, which would have an important clinical application in the health of this population, especially living in conditions of sedentarism and frailty in long-term institutions.

Aim: The present study analyzed the effects of twelve weeks of Capoeira training on the lipid profile of advanced-age frail adults of a long-term institution, which are characterized by sedentary lifestyle and affected by several diseases.

Methods: Participants were assigned into two groups (CONTROL: n = 07; 82.4±13.6 years and CAPOEIRA: n = 07; 79.4±6.9 years). The CAPOEIRA group performed twelve weeks of Capoeira training program, being twice a week lasting 60 minutes each at light to moderate intensity. Samples of 10 ml of blood were collected from participants' antecubital vein at the pre- and post-intervention moments in both groups. Plasma concentrations of triglycerides, total cholesterol, low density lipoprotein cholesterol and high density lipoprotein cholesterol were evaluated using the enzymatic colorimetric method. Anthropometry measures were performed and to internal control the energy consumption evaluations were carried out through daily food diaries during intervention period.

ELIGIBILITY:
Inclusion Criteria:

* age greater than 60 years;
* is not engaged in physical exercise programs for at least one year;
* do not present severe cardiovascular disease, kidney disease, liver disease or limiting cognitive or neuromuscular disease and;
* does not present visual or auditory inability.

Exclusion Criteria:

* failing to perform any of the evaluations suggested during the intervention protocol and;
* absence in five or more Capoeira training sessions.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-05-18 (Actual); Study Completion 2017-05-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline triglycerides concentration at 3 months | Pre- (week zero) and Post- (through study completion, 12 weeks) in Capoeira training group and Control group
  Samples of 10 ml of blood (to analyse triglycerides concentration in mg.dL-1) were collected from participants' antecubital vein from a 12-hour fast at the pre- and post-intervention moments of the CONTROL and CAPOEIRA groups.

CONTACTS AND LOCATIONS:
Overall Officials: Sérgio R Moreira, PhD, Principal Investigator — Federal University of Vale do São Francisco
Locations (1):
- Federal University of Vale do São Francisco (UNIVASF)., Petrolina, Pernambuco, Brazil

REFERENCES:
- [Background] Moreira SR, Teixeira-Araujo AA, Dos Santos AO, Simoes HG. Ten weeks of capoeira progressive training improved cardiovascular parameters in male practitioners. J Sports Med Phys Fitness. 2017 Mar;57(3):289-298. doi: 10.23736/S0022-4707.16.06030-8. Epub 2016 Feb 3. PMID 26842867
- [Background] Moreira SR, Teixeira-Araujo AA, Numata Filho ES, Moraes MR, Simoes HG. Psychophysiological characterization of different capoeira performances in experienced individuals: A randomized controlled trial. PLoS One. 2018 Nov 15;13(11):e0207276. doi: 10.1371/journal.pone.0207276. eCollection 2018. PMID 30440010
- [Background] Moreira SR, Carvalho FO, Moraes JFVN, Carvalho RGS, Araújo RC, Teixeira-Araújo AA, Okano AH. Eight weeks of Capoeira progressive training program increases flexibility of beginners. Sport Sci Health 12: 329-337, 2016.